CLINICAL TRIAL: NCT00937547
Title: Observational Study for Determine the Presence and Genotypes of HVP Infection in Cervical Intraepithelial Neoplasia Grade II-III (CIN II-III), and Stage I Cervical Epidermoid Carcinoma and Cervical Adenocarcinoma.
Brief Title: Human Papillomavirus Infection and Virus Genotyping in Uterine Cervix Cancer in Venezuela
Acronym: HPI
Status: Completed | Type: Observational
Sponsor: Instituto Oncologico Luis Razetti (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr. Jorge Sanchez Lander, Dr. Jorge Sanchez-Lander, Instituto Oncologico Luis Razetti
Other Study IDs: CERVICAL CANCER AND HPV
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Results first posted 2012-11-08 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; Human Papillomavirus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4.1. Collection of cervical samples:
  1. Previous ethics committe approval (Instituto Venezolano de Investigaciones Cientificas and Instituto de Oncología Luis Razetti), we are going to collect paraffin bloks of 300 patients with hystologic diagnosis of CIN 2/3 or Stage I cervical cancer.
  The samples will be obtained from archives of the Pathology Units of the following medical centers in Venezuela: Instituto de Oncología Luis Razetti, Anatomía Patológica Universidad Central de Venezuela, Hospital Oncológico Pérez Carreño (Valencia), Maracaibo, Barquisimeto, Ciudad Bolívar, Puerto La Cruz, Mérida and Barinas.
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Hypothesis:

   If high risk genotypes of human papillomavirus (HPV) is the cause of cervical cancer worldwide, the genotypes associated with cervical cancer in Venezuela would be the same types found in other countries.
2. Objectives:

Primary objective:

The objective of this investigation is to determine the presence and genotypes of HVP infection in cervical intraepithelial neoplasia grade 2/3 (CIN 2/3), and Stage I cervical epidermoid carcinoma and cervical adenocarcinoma.

Specific objectives:

To establish the presence of HPV in cervical cancer patients in Venezuela by geographic distribution.

To establish which HPV types are linked with cervical cancer in Venezuela by geographic distribution.

DETAILED DESCRIPTION:
In Venezuela, cervical cancer is the second leading cause of cancer mortality in women. In developed countries, although it is not the first cause of cancer mortality, occupies a remarkable place in the neoplastic pathology (Cannistra, 1996; Dey, 1998).

Human Papilloma Virus (HPV) is involved in the development of cervical cancer, specially oncogenic types 16 and 18 (Koskela, 2000; Markowska, 1999).

To date, it is still unknown which HPV types are more frequent in Venezuela. Several studies made in this country concluded that HPV 16 is the predominant type in cervical pathology (Graterol 2006, Correnti 1997, Muñoz 2003), but there has not been performed a HVP genotyping to detect all the types involved in patients with cervical cancer. Neither has been establish which HPV types are more frequently involved in genital warts in Venezuela.

The goal of this investigation is perform a genotypification of HPV in cervical cancer and cervical intraepithelial neoplasia 2 and 3 in Venezuela to determine which types are more frequently related to this disease in our country.

4. STUDY DESIGN:

4.1. Collection of cervical samples:

1. Previous ethics committee approval (Instituto Venezolano de Investigaciones Cientificas and Instituto de Oncología Luis Razetti), we are going to collect paraffin blocks of 300 patients with histological diagnosis of CIN 2-3 or Stage I cervical cancer.

The samples will be obtained from archives of the Pathology Units of the following medical centers in Venezuela: Instituto de Oncología Luis Razetti, Anatomía Patológica Universidad Central de Venezuela(Caracas), Hospital Oncológico Pérez Carreño (Valencia), Maracaibo, Barquisimeto, Ciudad Bolívar, Puerto La Cruz, Mérida and Barinas.

Inclusion criteria:

1. Paraffin blocks with CIN 2/3, and Stage I cervical cancer biopsies obtained between 2001 and 2011.
2. Properly blocks identification in order to obtain personal and clinical patient information.

4.2. Molecular biology procedures:

1. Histologically handling of tissue: previous identification of pathologic lesions as described in inclusion criteria by an expert pathologist (sample with lesion but without necrosis), the paraffin block will be cut into 5 to 7 µm slides with new blades and gloves for each cut. It will be obtain 1 slides that will be distributed as follows: one sample will be send to Laboratorio de Virología Molecular del Instituto Venezolano de Investigaciones Científicas; the remained sample will be kept for further evaluation if is necessary. Each slide will be placed in a proper container and will be identified by a serial number in order to preserve patient intimacy and avoid biased results.
2. Deparaffinisation as described in Coombs 1999.
3. Tissue digestion, DNA extraction and precipitation as described in Gravitt 2000.
4. HPV genotyping will be detected by INNOLiPA system. The results will be correlated with clinical information.

ELIGIBILITY:
Inclusion Criteria:

paraffin blocks of 329 patients with histologic diagnosis of CIN 2, CIN 3 or Stage I cervical cancer. -

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cervical samples
Sampling Method: Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge sanchez, MD, Principal Investigator — Instituto Oncologico Luis Razetti
Locations (2):
- Venezuela (2):
  - Instituto Oncologico Luis razetti, Caracas, DF
  - Jorge Sanchez Lander, Caracas, Miranda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Samples were collected from files between 2001-2011
Pre-assignment Details: 14 samples were excluded because of misdiagnosis.
Groups:
- Invasive Cervical Cancer: patients with histologic diagnosis invasive cervical cancer.
- Cervical Intraepithelial Neoplasia 2: patients with histological diagnosis of cervical intraepithelial neoplasia grade 2
- Cervical Intraepithelial Neoplasia 3: patients with histological diagnosis of cervical intraepithelial neoplasia grade 3
Period: Overall Study
Arm/Group | Invasive Cervical Cancer | Cervical Intraepithelial Neoplasia 2 | Cervical Intraepithelial Neoplasia 3
Started | 96 | 84 | 149
Histological Samples | 95 | 78 | 142
Completed | 95 | 78 | 142
Not Completed | 1 | 6 | 7
Not completed — misdiagnosis | 1 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Invasive Cervical Cancer: Paraffin-embedded samples with histological diagnosis of invasive cervical cancer
- Intraepithelial Cervical Neoplasia 3: Paraffin-embedded samples with histological diagnosis of cervical intraepithelial neoplasia grade 3
- Intraepithelial Cervical Neoplasia 2: Paraffin-embedded samples with histological diagnosis of cervical intraepithelial neoplasia grade 2
- Total: Total of all reporting groups
Arm/Group | Invasive Cervical Cancer | Intraepithelial Cervical Neoplasia 3 | Intraepithelial Cervical Neoplasia 2 | Total
Number analyzed (Participants) | 96 | 149 | 84 | 329
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 1 | 4
  Between 18 and 65 years | 90 | 146 | 81 | 317
  >=65 years | 4 | 2 | 2 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.04) | 37.6 (10.42) | 36.9 (9.34) | 39.27 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 149 | 84 | 329
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Venezuela | 96 | 149 | 84 | 329

OUTCOME MEASURES:

1. Primary Outcome: HPV Identification
Description: HPV distribution was identified in CIN2, CIN3 and invasive cervical cancer
Time Frame: 6 months
Measure: Number; unit: biopsies
Groups:
- Invasive Cervical Cancer: Paraffin-embedded sample with histological diagnosis of invasive cervical cancer
- Cervical Intraepithelial Neoplasia 3: Paraffin-embedded sample with histological diagnosis of cervical intraepithelial neoplasia grade 3
- Cervical Intraepithelial Neoplasia 2: Paraffin-embedded sample with histological diagnosis of cervical intraepithelial neoplasia grade 2
Arm/Group | Invasive Cervical Cancer | Cervical Intraepithelial Neoplasia 3 | Cervical Intraepithelial Neoplasia 2
Number analyzed (Participants) | 96 | 149 | 84
biopsies | 95 | 142 | 78

2. Primary Outcome: HPV Type 16
Description: Number of biopsies positive to HPV 16.
Time Frame: 6 months
Measure: Number; unit: biopsies
Arm/Group | Invasive Cervical Cancer | Cervical Intraepithelial Neoplasia 3 | Cervical Intraepithelial Neoplasia 2
Number analyzed (Participants) | 95 | 142 | 78
biopsies | 65 | 90 | 35

3. Primary Outcome: HPV Type 18
Description: Number of biopsies positive to HPV 18.
Time Frame: 6 months
Measure: Number; unit: biopsies
Arm/Group | Invasive Cervical Cancer | Cervical Intraepithelial Neoplasia 3 | Cervical Intraepithelial Neoplasia 2
Number analyzed (Participants) | 95 | 142 | 78
biopsies | 11 | 14 | 5

4. Primary Outcome: HPV Type 31
Description: Number of biopsies positive to HPV 31.
Time Frame: 6 months
Measure: Number; unit: biopsies
Arm/Group | Invasive Cervical Cancer | Cervical Intraepithelial Neoplasia 3 | Cervical Intraepithelial Neoplasia 2
Number analyzed (Participants) | 95 | 142 | 78
biopsies | 6 | 10 | 8

5. Primary Outcome: HPV Type 33
Description: Number of biopsies positive to HPV 33.
Time Frame: 6 months
Measure: Number; unit: biopsies
Arm/Group | Invasive Cervical Cancer | Cervical Intraepithelial Neoplasia 3 | Cervical Intraepithelial Neoplasia 2
Number analyzed (Participants) | 95 | 142 | 78
biopsies | 6 | 10 | 5

6. Primary Outcome: HPV Type 45
Description: Number of biopsies positive to HPV 45.
Time Frame: 6 months
Measure: Number; unit: biopsies
Arm/Group | Invasive Cervical Cancer | Cervical Intraepithelial Neoplasia 3 | Cervical Intraepithelial Neoplasia 2
Number analyzed (Participants) | 95 | 142 | 78
biopsies | 6 | 6 | 5

7. Primary Outcome: HPV Type 58
Description: Number of biopsies positive to HPV 58.
Time Frame: 6 months
Measure: Number; unit: biopsies
Arm/Group | Invasive Cervical Cancer | Cervical Intraepithelial Neoplasia 3 | Cervical Intraepithelial Neoplasia 2
Number analyzed (Participants) | 95 | 142 | 78
biopsies | 3 | 7 | 5

8. Primary Outcome: HPV Type 51
Description: Number of biopsies positive to HPV 51.
Time Frame: 6 months
Measure: Number; unit: biopsies
Arm/Group | Invasive Cervical Cancer | Cervical Intraepithelial Neoplasia 3 | Cervical Intraepithelial Neoplasia 2
Number analyzed (Participants) | 95 | 142 | 78
biopsies | 1 | 5 | 7

ADVERSE EVENTS:
Description: No adverse event assessment because there were no patient intervention, there were used biopsies from archives for the analysis.
Arm/Group | Invasive Cervical Cancer | Intraepithelial Cervical Neoplasia 3 | Intraepithelial Cervical Neoplasia 2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No